CLINICAL TRIAL: NCT04397770
Title: Camrelizumab Plus Apatinib and Temozolomide as First Line Therapy in Advanced Acral Melanoma：a Single-center, Exploratory Clinical Study
Brief Title: Camrelizumab Plus Apatinib and Temozolomide as First Line Therapy in Advanced Acral Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jun Guo, Associate Director of Peking University Cancer Hospital, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-MM-II-002
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — camrelizumab; apatinib; Temozolomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camre+Apa+TMZ (Experimental)
  Interventions: Drug: SHR1210; Drug: apatinib mesylate; Drug: Temozolomide Injection

INTERVENTIONS:
Drug: SHR1210 — SHR-1210 is a humanized anti-PD1 IgG4 monoclonal antibody
Drug: apatinib mesylate — apatinib Mesylate is a small molecule tyrosine kinase inhibitor,Through selectively inhibiting the tyrosine kinase activity of the vascular endothelial growth factor receptor 2 (VEGFR-2).
Drug: Temozolomide Injection — Temozolomide is an imidazole tetrazine derivative of the alkylating agent dacarbazine.Temozolomide is not directly active but undergoes rapid, spontaneous, non-enzymatic conversion at physiologic pH to the cytotoxic compound, monomethyl triazeno imidazole carboxamide (MTIC).

SUMMARY:
It is a single-center,exploratory clinical trial aimed to evaluate the objective response rate (ORR) of Camrelizumab combined with apatinib and Temozolomide as First Line Therapy in Advanced Acral Melanoma.

ELIGIBILITY:
Inclusion Criteria:

1. age:18-75 years, male or female.
2. Histopathologically confirmed recurrence, inoperable resection or metastatic acral melanoma (stage III/IV).
3. Has not received any systematic anti-tumor drug treatment.
4. Measurable disease based on Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.
5. ECOG 0-1.
6. Adequate organ function.
7. Life expectancy of greater than 12 weeks.
8. Patient has given written informed consent.

Exclusion Criteria:

1. Patients who have or are currently undergoing additional chemotherapy, radiation therapy, targeted therapy or immunotherapy.
2. Known history of hypersensitivity to macromolecular protein preparation or any components of the SHR- 1210 formulation.
3. Subjects before or at the same time with other malignant tumors (except which has cured skin basal cell carcinoma and cervical carcinoma in situ);
4. Subjects with any active autoimmune disease or history of autoimmune disease
5. Uncontrolled clinically significant heart disease, including but not limited to the following: (1) > NYHA II congestive heart failure; (2) unstable angina, (3) myocardial infarction within the past 1 year; (4) clinically significant supraventricular arrhythmia or ventricular arrhythmia requirement for treatment or intervention;
6. Active infection or an unexplained fever > 38.5°C during screening or before the first scheduled day of dosing (subjects with tumor fever may be enrolled at the discretion of the investigator);
7. Received a live vaccine within 4 weeks of the first dose of study medication.
8. Pregnancy or breast feeding.
9. Decision of unsuitableness by principal investigator or physician-in charge.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
ORR | Through study uncompletion, an average of 1 year
  Objective Response Rate

REFERENCES:
- [Derived] Mao L, Lian B, Li C, Bai X, Zhou L, Cui C, Chi Z, Sheng X, Wang X, Tang B, Yan X, Li S, Kong Y, Dai J, Wei X, Li J, Duan R, Xu H, Wu X, Yang Y, Cheng F, Zhang C, Xia F, Pang Z, Guo J, Si L. Camrelizumab Plus Apatinib and Temozolomide as First-Line Treatment in Patients With Advanced Acral Melanoma: The CAP 03 Phase 2 Nonrandomized Clinical Trial. JAMA Oncol. 2023 Aug 1;9(8):1099-1107. doi: 10.1001/jamaoncol.2023.1363. PMID 37261804